CLINICAL TRIAL: NCT01748578
Title: A Phase 1, Double-Masked, Placebo-Controlled, Dose Escalating Study of the Safety, Tolerability, and Pharmacokinetics of EBI-005 Topically Administered to Eyes of Healthy Adult Subjects
Brief Title: Phase 1 Study for Safety and Tolerability of EBI-005 Topically Administered to Eyes of Healthy Adult Subjects
Acronym: EBI-005-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eleven Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBI-005-1
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Dry Eye
Keywords: Healthy; Interleukin 1 Receptor Inhibitor; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBI-005-1 5mg/mL (Active Comparator): Healthy subjects will be randomized to EBI-005 5mg/mL vs. EBI-005-1 Placebo 3x/day
  Interventions: Drug: EBI-005-1; Drug: EBI-005-1 Placebo
- EBI-005-1 20 mg/mL (Active Comparator): Healthy subjects will be randomized to EBI-005 20 mg/mL vs. EBI-005-1 Placebo 3x/day
  Interventions: Drug: EBI-005-1; Drug: EBI-005-1 Placebo

INTERVENTIONS:
Drug: EBI-005-1 — EBI-005-1 is an intervention to two different study arms: 5mg/ml Vs Placebo and 20 mg/ml Vs Placebo
Drug: EBI-005-1 Placebo

SUMMARY:
This is a First-In-Human (FIH) study to assess the safety and tolerability of ocular administration of EBI-005 in healthy volunteers. Additionally, the PK and immunogenicity of EBI-005 will be assessed.

DETAILED DESCRIPTION:
The planned dose levels are 5 mg/mL EBI-005 (Group 1) and 20 mg/mL EBI-005 (Group 2).

A total of 8 subjects will be dosed in each group with subjects randomized in a ratio of 6:2, EBI-005:placebo. Treatment administration in Group 2 will proceed following a review of safety data from Group 1. In both groups, subjects randomized to active treatment will receive EBI-005 in the right eye and placebo in the left eye. Subjects randomized to placebo will receive placebo in each eye.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females between the ages of 18 and 65 years
* Medically healthy
* Best correction vision of greater than or equal to 20/40 in each eye
* Non-tobacco/nicotine-containing product users for a minimum of 6 months prior to dosing
* Tolerate topical administration to eye
* Signed and dated, Institutional Review Board (IRB) approved informed consent form (ICF) prior to any protocol-specific screening procedures

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic (including sensitive skin on the face), neurological, or psychiatric disease, or any other clinically significant disease not deemed acceptable by the PI
* History of any primary malignancy, with the exception of basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ or other malignancies curatively treated and with no evidence of disease for at least 5 years
* Occurrence of active seasonal allergies including ocular allergies (e.g.; annual hay fever)
* Abnormalities following ophthalmological examination: abnormality of the cornea, evidence of ocular inflammation (dry eyes, blepharitis, allergic conjunctivitis, iritis, and uveitis), glaucoma, and optic neuropathy
* Subjects with a history of laser refractive surgery (laser assisted stromal in-situ keratomileusis [LASIK], photorefractive keratectomy [PRK]), radial keratotomy (RK), corneal transplantation, dry eyes, or radiotherapy to the eyes
* Use of contact lenses currently or within the past one year
* Positive urine drug/alcohol or cotinine testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in ocular safety measurements. | 1 week
  Determined by best corrected visual acuity, slit lamp examination, measurement of intraocularpressure (IOP)

SECONDARY OUTCOMES:
ELISA based assay to determine Pharmacokinetics for the evaluation of systemic exposure of EBI-005 in healthy volunteers. | 1 week
ELISA based assay to determine Immunogenicity for the evaluation of systemic exposure of EBI-005 in healthy volunteers. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldstein, MD, Study Director — Eleven Biotherapeutics
Locations (1):
- Celerion, Tempe, Arizona, United States